CLINICAL TRIAL: NCT00905866
Title: Evaluation of Quality of Life in Patients Undergoing Parathyroidectomy
Brief Title: Quality of Life in Patients Undergoing Parathyroidectomy
Status: Completed | Type: Observational
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Shih-Ping Cheng, MD, Mackay Memorial Hospital
Other Study IDs: MMH-I-S-591
Record Dates: First submitted 2009-05-18; First posted 2009-05-21 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Parathyroidectomy; Hyperparathyroidism
Keywords: Quality of life; Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Quality of life: All participants undergoing parathyroidectomy
  Interventions: Other: PAS and SF-36 questionnaires

INTERVENTIONS:
Other: PAS and SF-36 questionnaires — Patients who agree to participate in this study will be asked to fill out a translated PAS questionnaire and a Taiwan version of SF-36 before and after surgery

SUMMARY:
There are three specific aims in the present study:

1. To validate the investigators' translated version of parathyroidectomy assessment of symptoms (PAS) questionnaire.
2. To evaluate the impact of parathyroidectomy on health-related quality of life in the investigators' patients with hyperparathyroidism.
3. To analyze the association between clinical variables and the presentation/severity of symptoms (and/or quality of life domains) in the investigators' patients.

DETAILED DESCRIPTION:
Either primary or secondary hyperparathyroidism may necessitate parathyroidectomy in some patients to improve the related biochemical abnormalities or symptoms, or both. Many patients diagnosed with hyperparathyroidism today do not have the classic or historical severe manifestations such as osteitis fibrosa cystica or nephrocalcinosis. The well-known pentad of symptoms - painful bones, kidney stones, abdominal groans, psychic moans, and fatigue overtones - is more common, although most patients have few dramatic symptoms. The multifactorial causes for many of the symptoms that patients have make it difficult to know to what extent surgical intervention will alleviate the symptoms. Several endocrine surgeons from the western countries have used a standardized health status assessment tool such as the SF-36 (the Medical Outcomes Study Short-Form Health Survey) to assess symptoms and health state in patients with hyperparathyroidism. Results of the studies confirmed that these patients are indeed impaired in several domains and even seemingly "asymptomatic" patients benefit from parathyroidectomy. More recently, Canadian surgeon Pasieka designed and validated a disease-specific surgical outcome tool, the parathyroidectomy assessment of symptoms (PAS) score, for patients with hyperparathyroidism. Using this tool, several studies from different countries showed that the study group of patients with hyperparathyroidism had significantly more symptoms than controls, and some of the symptoms are remarkably ameliorated after surgery. In Taiwan, only a small number of studies have evaluated neuropsychiatric function and neuromuscular abnormalities in these patients. None of the studies has used a patient-based measure of health status or quality of life intended to capture patient-reported perceptions of health and function.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and older

Exclusion Criteria:

* Subjects who are illiterate or unable to complete questionnaire
* Excluded by patient's clinician prior to recruitment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients underwent parathyroidectomy
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2008-08; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the impact of parathyroidectomy on health-related quality of life in patients with hyperparathyroidism | 1 year

SECONDARY OUTCOMES:
To analyze the association between clinical variables and the presentation/severity of symptoms (and/or quality of life domains) in patients undergoing parathyroidectomy | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Ping Cheng, MD, Principal Investigator — Mackay Memorial Hospital
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Adler JT, Sippel RS, Schaefer S, Chen H. Surgery improves quality of life in patients with "mild" hyperparathyroidism. Am J Surg. 2009 Mar;197(3):284-90. doi: 10.1016/j.amjsurg.2008.09.009. PMID 19245902
- [Background] Pasieka JL, Parsons LL, Demeure MJ, Wilson S, Malycha P, Jones J, Krzywda B. Patient-based surgical outcome tool demonstrating alleviation of symptoms following parathyroidectomy in patients with primary hyperparathyroidism. World J Surg. 2002 Aug;26(8):942-9. doi: 10.1007/s00268-002-6623-y. Epub 2002 May 21. PMID 12016473
- [Background] Pasieka JL, Parsons LL. A prospective surgical outcome study assessing the impact of parathyroidectomy on symptoms in patients with secondary and tertiary hyperparathyroidism. Surgery. 2000 Oct;128(4):531-9. doi: 10.1067/msy.2000.108117. PMID 11015085
- [Background] Greutelaers B, Kullen K, Kollias J, Bochner M, Roberts A, Wittert G, Pasieka J, Malycha P. Pasieka Illness Questionnaire: its value in primary hyperparathyroidism. ANZ J Surg. 2004 Mar;74(3):112-5. doi: 10.1111/j.1445-2197.2004.02907.x. PMID 14996155
- [Background] Chow KM, Szeto CC, Kum LC, Kwan BC, Fung TM, Wong TY, Leung CB, Li PK. Improved health-related quality of life and left ventricular hypertrophy among dialysis patients treated with parathyroidectomy. J Nephrol. 2003 Nov-Dec;16(6):878-85. PMID 14736016
- [Background] Cheng SP, Liu CL, Chen HH, Lee JJ, Liu TP, Yang TL. Prolonged hospital stay after parathyroidectomy for secondary hyperparathyroidism. World J Surg. 2009 Jan;33(1):72-9. doi: 10.1007/s00268-008-9787-2. PMID 18953601